CLINICAL TRIAL: NCT04766151
Title: A Randomised, Double-blind, Parallel Group, Efficacy and Safety Study of Transdermal Patch Nitroglycerin in the Prevention of Coronary Artery Spasm, During Coronary Angiography/ Angioplasty (NURSE-TTS - Nitrate Use to Obtain Radial Spasm Embarrassment)
Brief Title: Nitrate Use to Obtain Radial Spasm Embarrassment (NURSE - TTS Trial)
Acronym: NURSE-TTS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: 424 General Military Hospital (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Fotios Oikonomou, Consultant Interventional Cardiologist - Head of Cath Lab, 424 General Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 27
Record Dates: First submitted 2021-02-15; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Radial Artery Spasm
MeSH Terms: interventions — Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transdermal glyceryl trinitrate patches (Experimental)
  Interventions: Drug: Transdermal glyceryl trinitrate 10mg patches
- Transdermal placebo patches (Placebo Comparator)
  Interventions: Drug: Placebo patches

INTERVENTIONS:
Drug: Transdermal glyceryl trinitrate 10mg patches — Transdermal patches applied to skin 30 minutes before cardiac catheterization
  Other Names: Nitrong tts 10mg- Lavipharm S.A.
  Arms: Transdermal glyceryl trinitrate patches
Drug: Placebo patches — Transdermal placebo patches applied to skin 30 minutes before cardiac catheterization
  Arms: Transdermal placebo patches

SUMMARY:
Transradial cardiac catheterization and percutaneous coronary intervention are increasingly being performed worldwide in elective and emergency procedures, with many centres adopting the transradial route as their first choice of arterial access. One of the most common complications encountered during transradial procedures is radial artery spasm. The aim of this study is to evaluate the Efficacy and Safety of the use of transdermal Glyceryl trinitrate patches applied to skin before cardiac catheterization to prevent the occurrence of radial artery spasm during transradial access cardiac catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 -85 years old who has been admitted for scheduled coronary angiography by radial artery

Exclusion Criteria:

* Prior same radial artery catheterization
* Positive Allen test
* Severe Hypotension (SBP<100 mmHg)
* Pregnancy
* Ongoing Acute Myocardial Infarction
* Ongoing cardiogenic shock
* Known History of Nitrates intolerance/allergy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Radial Spasm occurrence | Immediately after the end of the procedure
  Radial spasm is measured by the exerting force (in Newton) removing the sheath from the patient
Successful radial puncture | During radial puncture and catheterization
  The success is defined by the fast radial puncture and catheterization and is measured by the time of radial catheterization

SECONDARY OUTCOMES:
VRS-4 pain scale | During the whole procedure
  The pain during the procedure is measured by the four-category verbal rating scale (VRS-4)
State-Trait Anxiety Inventory (STAI) | During the whole procedure
  The anxiety during the procedure is measured by the State - Trait Anxiety Inventory (STAI)

CONTACTS AND LOCATIONS:
Locations (1):
- 424 GeneralMH, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Economou FI, Doundoulakis I, Kalamakidou I, Koliastasis L, Soulaidopoulos S, Samara M, Dimitriadis K, Papazisis G, Tsiachris D, Tsioufis K. Prevention of Radial Artery Spasm With Transdermal Glyceryl Trinitrate Patches: The NURSE-TTS Randomized Study. JACC Cardiovasc Interv. 2023 Feb 13;16(3):365-367. doi: 10.1016/j.jcin.2022.09.032. Epub 2023 Jan 4. No abstract available. PMID 36609046